CLINICAL TRIAL: NCT03703076
Title: A Post-Authorisation Non-Interventional Observational, Multi-Site Study of Patients in France With Primary Biliary Cholangitis Treated With Obeticholic Acid in Real Life (OCARELIFE)
Brief Title: A Post-Authorisation Non-Interventional Observational of Patients in France With Primary Biliary Cholangitis Treated With Obeticholic Acid in Real Life
Acronym: OCARELIFE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: SAMEY (Industry)
Collaborators: Axonal-Biostatem (Industry)
Responsible Party: Sponsor-Investigator, SAMEY, CRO Project manager, Intercept Pharma France SAS
Organization: Intercept Pharma France SAS (Industry)
Other Study IDs: 2018-A00075-50
Record Dates: First submitted 2018-10-09; First posted 2018-10-11 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Post-authorisation non-interventional observational study of patients with Primary Biliary Cholangitis who started Ocaliva® treatment between October 1st, 2016 and December 31, 2017.

DETAILED DESCRIPTION:
This is a non-interventional, multi-site, ambispective, national follow-up study of patients with Primary Biliary Cholangitis who started Ocaliva® treatment between October 1st, 2016 and December 31, 2017. This represents approximately 150 patients to date, who are therefore the first patients to have received treatment with Ocaliva® in France outside of pre-approval clinical trials.

All patients who received treatment within the context of the ATU (conditional marketing authorization in France) or after EU marketing authorization approval for the product will be followed up for 18 months (this follow-up will be partly retrospective and partly prospective). The study therefore involves retrospective recruitment with retrospective and prospective data collection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PBC treated with Ocaliva® 5 mg or 10 mg according to the terms of Ocaliva® approved SmPC: in combination with ursodeoxycholic acid (UDCA) in adults with an inadequate response to UDCA or as monotherapy in adults unable to tolerate UDCA (over the age of 18 years at the time of treatment introduction).
* Patients with PBC with a suboptimal response to UDCA who received at least one dose of Ocaliva®.
* Patients with or without an overlap syndrome (Nguyen-Khac E, 2004)
* Prior to any follow-up and inclusion in this cohort, the attending physician must give the patient or his or her legal representative or designated healthcare proxy information on the drug, a side effect report and notice of his or her inclusion in the cohort (patient information sheet in writing).
* The patient (or his or her legal representative or designated healthcare proxy) must have read the information sheet and agreed verbally to take part, and must show the sheet to any doctor who is consulted.

Exclusion Criteria:

* Diseases triggering a non-hepatic elevation of alkaline phosphatases (ALP) (for example Paget's disease or fractures within the previous three months).
* Participation in another investigational study on a product, biological material or medical device within the 30 days prior to selection.
* Inability to comply with the study follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients with PBC treated between October 1st, 2016 and December 31, 2017 with Ocaliva® 5 mg or 10 mg according to the terms of Ocaliva® approved SmPC: in combination with ursodeoxycholic acid (UDCA) in adults with an inadequate response to UDCA or as monotherapy in adults unable to tolerate UDCA (over the age of 18 years at the time of treatment introduction).
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-04-10 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Response to Ocaliva® after 12 months of treatment | 12 month
  Response to Ocaliva® after 12 months of treatment as monotherapy or in combination, using the published Paris 2 response criteria

SECONDARY OUTCOMES:
Response rate using the Paris 2 criteria at the end of the study | 18 month
  Response rate using the Paris 2 criteria at the end of the study, 18 month after treatment initiation

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Chu Grenoble, Grenoble
  - Hopital Saint Antoine, Paris